CLINICAL TRIAL: NCT03704363
Title: The Effect of Infliximab in Patients With Chronic Low Back Pain and Modic Changes. A Randomized, Double Blind, Placebo-controlled, Multicenter Trial
Brief Title: BackToBasic: Infliximab in Chronic Low Back Pain and Modic Changes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Haukeland University Hospital (Other); St. Olavs Hospital (Other); University Hospital of North Norway (Other); Vestre Viken Hospital Trust (Other); Ostfold Hospital Trust (Other); Clinical Trial Unit (CTU), Oslo University Hospital (Unknown); Diakonhjemmet Hospital (Other)
Responsible Party: Principal Investigator, Kjersti Storheim, Oslo University Hospital, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017/2450
Record Dates: First submitted 2018-09-19; First posted 2018-10-12 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Low Back Pain
Keywords: Modic changes; biomarkers; treatment; infliximab; chronic low back pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A computer-generated randomised allocation sequence will be imported into an electronic case report form (eCRF) system (Viedoc) and made available exclusively to a study nurse (mixing nurse) authorised by the local principal investigator to prepare infusions. The mixing nurse is otherwise not involved in the treatment of the patient. The infusion bags containing the study medication will be prepared by the mixing nurse in identical infusion bags, and applied labels with patient number and dose such that blinding of the participants is secured. The Investigational Medicinal Products (IMPs) have the same color and will look the same. After preparing the IMP, the mixing nurse will hand over the IMP to another nurse, blinded to allocation, and authorised by the local principal investigator to administer the infusion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Infliximab (Experimental): Intravenous infusion(biosimilar infliximab). Each participant will be given 4 infusions, at day 0, day 14, day 42 and day 98, unless unacceptable toxicity is encountered.
  Interventions: Drug: Biosimilar Infliximab
- Placebo (Placebo Comparator): Intravenous infusion (NaCl intravenous infusion). Each participant will be given 4 infusions, at day 0, day 14, day 42 and day 98.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Biosimilar Infliximab — Intravenous infusion(5 mg/kg). Each participant will be given 4 infusions, at day 0, day 14, day 42 and day 98, unless unacceptable toxicity is encountered.
  Arms: Infliximab
Other: Placebo — Intravenous infusion. Each participant will be given 4 infusions, at day 0, day 14, day 42 and day 98,
  Other Names: NaCl intravenous infusion
  Arms: Placebo

SUMMARY:
Low-Back Pain (LBP) is the leading cause of disability worldwide. Even though LBP relates to different underlying pathologies, there are a substantial number of patients with chronic complaints that have vertebral bone marrow lesions visualized as Modic changes (MC) on magnetic resonance imaging (MRI). Despite the clinical evidence that MC is painful, the etiology is unknown and there is currently no established treatment. It has been suggested that MCs are secondary to a biomechanically induced degradation with a subsequent autoimmune response, supported by evidence showing that Tumor necrosis factor (TNF)-α plays a critical role in intervertebral disc degeneration and MCs. Clinical trials suppressing inflammation with TNF-alfa blockers in patients with acute low back pain and sciatica provide evidence to support the initiation of a clinical trial assessing the effect of TNF-alfa blockers in patients with chronic low-back pain and MCs. Since TNF-alfa blockers is an established treatment for immune-mediated disorders like spondyloarthritis by reducing pain as well as bone marrow lesions, the researchers aim to assess whether this treatment is effective for chronic LBP with MCs. In addition refine diagnostic assessment and explore potential biomarkers, which will provide an increased understanding of underlying factors causing LBP, and ultimately result in better management and treatment for one of the most costly and challenging patient populations.

DETAILED DESCRIPTION:
The following information will be collected at baseline, in addition to pre-specified efficacy assessments: age, gender, BMI (measured at site), ethnicity, marital status, children, educational level, work status, physical work load, leisure time activity, smoking habits, expectations about treatment effect and characteristics of pain (duration, agrevating factors, morning stiffness, morning pain, relief by NSAIDs, night time pain and former treatment). Emotional distress will be measured using the Hopkins Symptom Checklist-25 at baseline. The researchers will measure fear-avoidance beliefs about physical activity and work with Fear-avoidance beliefs Questionnaire (FABQ) at baseline. Subjective health complaints (SHC) will be measured using a formal inventory which consists of 29 questions concerning severity and duration of subjective somatic and psychological complaints and will be measured at baseline. In addition, routine clinical investigations (pain provocation tests (springing test, active flexion / extension of the lumbar spine) and neurological tests (strength, toe-/heel walking, sensibility, reflexes, straight leg raising test, reverse Lasegue test)) will be structured and registered in the CRF at baseline.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* LBP of > 50% of days for > 6 months duration in the area below the 12th rib and above the gluteal folds with:

Numerical Rating Scale (NRS) pain intensity score of at least 5 (mean of three NRS scales; current LBP, the worst LBP within the last 2 weeks, and usual/mean LBP within the last 2 weeks) and/or ODI-score of at least 25

- Modic change of craniocaudal size >= 10% of vertebral height and of primary or secondary type 1 in the vertebral body at a level of the lumbar spine (superior or inferior endplate, Th12-S1).

Exclusion criteria:

* Fever or ongoing infection
* Allergy or hypersensitivity against any products of the medication
* Previous infliximab treatment
* Any serious adverse events with other immunosuppressive treatment (including cytostatics, antibodies, drugs acting on immunophilins, Interferons, mycophenolate and any other DMARDs)
* Any specific diagnosis that may explain patient's low back symptoms (e.g. tumor, fracture, spondyloarthritis, infection, spinal stenosis).
* Former low back surgery (L1 - S1) for other reasons than disc herniation or decompression (e.g fusion, disc prosthesis).
* Former surgery for disc herniation or decompression within the last 12 months
* Any known rheumatic disease
* Current pregnancy or lactation
* For women of childbearing potential (WOCBP); inadequate birth control, pregnancy, and/or breastfeeding. WOCBP is defined as those who are fertile (with uterus, fallopian tubes and at least one intact functional ovary), following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy. Documentation of surgical procedure or physical examination is required for subjects who have had such an operation. Adequate contraception must be used by WOCBP during the entire intervention period and 6 months after the last administration of study drug, and includes oral, injected or implanted hormonal methods of contraception, placement of an intrauterine device or system, vasectomized partner or sexual abstinence.
* Ongoing systemic glucocorticoid or other immunosuppressive treatments (see list above)
* Regular use of opioids with the exception of codeine and tramadol
* Other immunosuppressive treatment last year (see list above)
* Active or latent (known or suspected) tuberculosis (all participants will be screened for latent tuberculosis)
* Previous infection with Hepatitis B virus (HBV) (all participants will be screened for HBV-carrier state)
* Live vaccination within the last 4 weeks or planned live vaccination during treatment period
* Planned surgical procedure
* Increased transaminases (ASAT/ALAT)
* Ongoing or previous malignant disease at any time (i.e. skin cancer, cervical cancer etc.)
* Known increased risk of malignant disease
* Diabetes
* Immunodeficiency (I.e primary immunodeficiency diseases, human immunodeficiency virus/acquired immunodeficiency syndrome, splenectomy)
* Heart failure (NYHA class III - IV)
* Previous or ongoing psoriasis
* Ulcerative colitis or Crohns disease
* Existing or recent demyelination diseases (I.e. MS or Guillain-Barres)
* Abnormal hemoglobin or abnormal platelet, leucocyte or neutrophil count
* Not able to understand written and spoken Norwegian
* Not able to complete treatment or follow-ups in the study (i.e. severe psychiatric disease, drug abuse or plans of moving address)
* Contraindications for MRI (ie. pacemaker, metal implants, claustrophobia)
* Abnormal creatinine level

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2023-07-27 (Actual); Study Completion 2023-09-29 (Actual)

PRIMARY OUTCOMES:
Change in Oswestry Disability Index (ODI) from baseline to 5 months | 0, 1, 2, 3, 4, 5 and 9 months
  ODI is a disease-specific disability score. Scale is measured 0-100, better to worse respectively.

SECONDARY OUTCOMES:
Change in Short tau inversion recovery (STIR) signal (intensity and extent) of Modic Changes from baseline to 5 months. | 0 and 5-6 months
  Based on Magnetic Resonance Imaging (MRI). STIR result from evaluations of fat-water separation and T1 weighted fat-saturated post-contrast images, MC signal intensity standardized against the intensity of normal vertebral body marrow and cerebrospinal fluid, MC high signal craniocaudal size and volume.
Change in low back pain intensity from baseline to 5 months | 0 + weekly during intervention period, 3, 5 and 9 months
  Measured on a Numeric Rating Scale (NRS: 0-10); mean of three NRS scales; current LBP, the worst LBP within the last 2 weeks, and usual/mean LBP within the last 2 weeks (at baseline, post-treatment and at one year after start of treatment). Will also be monitored weekly during the intervention period, and the the wording "last 2 weeks" will then be replaced by "the last week". Better (0) to worse (10) respectively.
Change in Roland Morris Disability Questionnaire (RMDQ) from baseline to 5 months | 0, 3, 5 and 9 months
  RMDQ is a Self-reported disease-specific disability score, scale 0-24, better to worse respectively.
Change in Health-related quality of life from baseline to 5 months | 0, 3, 5 and 9 months
  EuroQoL-5D-5L (version 2.0), range -0.59 to 1.0, worse to better respectively.
Number and type of co-interventions (other pharmacological treatment (ATC-coded) and non-pharmacological treatment) | Will be registered every month up to 5 months and at 9 months
  Will be reported by patients monthly during the study period for health-economical calculations
Days with sick leave | Will be registered at baseline and monthly until last follow-up
  Self-reported by patients; how many days patients were on sick-leave last month (if patients are sick listed; degree / % sick listed will also be registered).
Incidence of adverse events (AEs) and serious AE (SAEs) during the study period | 2, 6, 14, 22 and 40 weeks after start of treatment
  Adverse events frequency. The nature of the event(s) will be described by the investigator in precise standard medical terminology, duration and intensity will also be registered. In the evaluation, we will also consider serum infliximab concentration and vital signs.

OTHER OUTCOMES:
Change in Leg pain intensity from baseline to 5 months | 0, 3, 5 and 9 months
  Numeric Rating Scale (NRS: 0-10, better to worse respectively); leg pain last week.
Change in Hours with low back pain during the last 4 weeks from baseline to 5 months | 0, 3, 5 and 9 months
  Number of days during the last 28 days (4 weeks) the participant had experienced LBP (0-28 days), and, on an typical day, how many of the hours awake they experienced LBP (0-16 h). The number of days and hours are multiplied (a 0-448 scale).
Change in Symptom-specific well-being from baseline to 5 months | 0, 3, 5 and 9 months
  Measured on a 5-point Likert scale with 'very satisfied', 'some satisfied', 'neither satisfied nor dissatisfied', 'some dissatisfied' or 'very dissatisfied'
Patients' satisfaction | Will be measured at 3, 5 and 9 months after start of treatment
  Rated on a 5-point Likert scale; patients rate satisfaction with treatment
Global perceived effect from baseline | Will be measured at 3, 5 and 9 months after start of treatment
  Global Rating of Change is rated on a 7-point Likert scale to quantify a patient's self-judged improvement from baseline.
Perceived treatment | Seven days after start of treatment, post-treatment (14 weeks after start of treatment) and at 5 months after start of treatment
  Patients will be asked about which study medicine (Infliximab / placebo / unsure) they think they received during the intervention period of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Froholdt, PhD, Principal Investigator — Vestre Viken Hospital Trust Drammen; Anne Julsrud Haugen, PhD, Principal Investigator — Ostfold Hospital Trust; Jan Sture Skouen, PhD, Principal Investigator — Haukeland University Hospital; Jens Ivar Brox, PhD, Principal Investigator — Oslo University Hospital; Gunn Hege Marchand, PhD, Principal Investigator — St. Olavs Hospital, Trondheim; Gunnstein Bakland, PhD, Principal Investigator — University Hospital of North Norway Tromsø; John-Anker Zwart, PhD, Study Chair — Oslo University Hospital, Oslo, Norway
Locations (6):
- Norway (6):
  - Haukeland University Hospital, Bergen
  - Vestre Viken Hospital Trust Drammen, Drammen
  - Østfold Hospital Trust, Moss
  - Oslo University Hospital Ullevål, Oslo
  - University Hospital of North Norway, Tromsø
  - St. Olavs Hospital, Trondheim

REFERENCES:
- [Derived] Gjefsen E, Braten LCH, Goll GL, Wigemyr M, Bolstad N, Valberg M, Schistad EI, Marchand GH, Granviken F, Selmer KK, Froholdt A, Haugen AJ, Dagestad MH, Vetti N, Bakland G, Lie BA, Haavardsholm EA, Nilsen AT, Holmgard TE, Kadar TI, Kvien T, Skouen JS, Grovle L, Brox JI, Espeland A, Storheim K, Zwart JA. The effect of infliximab in patients with chronic low back pain and Modic changes (the BackToBasic study): study protocol of a randomized, double blind, placebo-controlled, multicenter trial. BMC Musculoskelet Disord. 2020 Oct 21;21(1):698. doi: 10.1186/s12891-020-03720-5. PMID 33087100

DOCUMENTS (2):
  • Statistical Analysis Plan: SAP for main clinical outcomes (2023-09-27): https://cdn.clinicaltrials.gov/large-docs/63/NCT03704363/SAP_000.pdf
  • Statistical Analysis Plan: SAP for MRI studies in BackToBasic (2024-03-04): https://cdn.clinicaltrials.gov/large-docs/63/NCT03704363/SAP_001.pdf